CLINICAL TRIAL: NCT06930469
Title: Application of Structured Team Model Based on Shared Decision Model in Obstetrics and Gynecology Joint Intensive Care Unit (ICU) Rescue of Critical Care Pregnant Women
Brief Title: Shared Decision-Making Structured Team Model for Critical Maternal Care in OB-GYN ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ying Wang (Other)
Responsible Party: Sponsor-Investigator, Ying Wang, Clinical Professor, Nantong First People's Hospital
Organization: Nantong First People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022KT096
Record Dates: First submitted 2025-03-25; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness; Pregnant Women
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- structured team model with shared decision-making (Experimental)
  Interventions: Behavioral: structured team model with shared decision-making
- conventional multidisciplinary resuscitation care (Other)
  Interventions: Behavioral: conventional multidisciplinary resuscitation care

INTERVENTIONS:
Behavioral: structured team model with shared decision-making — Structured team model based on shared decision-making model: ① Maternal Critical Care Review: Pre-hospital (prenatal checkup): Obstetricians and nurses conduct regular prenatal checkups for mothers, identify high-risk mothers, and set up high-risk maternal health records. Referral: Critically ill pregnant women establish a green channel for timely referral to the obstetrics department or ICU, and contact the relevant personnel of the structured management team. Assessment: The multidisciplinary team conducts a comprehensive assessment of the extent of the maternal condition, vital signs, and laboratory test results. Identification: Identify the main causes of critical maternal illness and potential risks, such as hemorrhage, infection, and organ failure. Rescue plan: according to the assessment results, formulate a personalized rescue plan and clarify the responsibilities and tasks of each department. Monitoring: real-time monitoring of maternal vital signs and changes in condition, a
  Arms: structured team model with shared decision-making
Behavioral: conventional multidisciplinary resuscitation care — The observation group implemented a structured team model based on a shared decision-making model, which operated as follows:
  (1) Constructing a structured management team: multidisciplinary medical and nursing staff, including obstetricians, ICU doctors, obstetric nurses, ICU nurses, head nurses, anesthesiologists, ultrasonographers, and family members of the patient's main companions, are divided into small teams according to their functions, and each small team has a team leader who is responsible for the coordination of the overall situation and the rapid coordination of information. Obstetricians and ICU doctors are responsible for life support, obstetric evaluation, condition monitoring and development of resuscitation plan for critically ill mothers. Anesthesiologists are responsible for anesthesia management, pain control and intraoperative resuscitation support. The nurse manager coordinates the nursing team to ensure the standardization of rescue care. Obstetrician and ICU nu
  Arms: conventional multidisciplinary resuscitation care

SUMMARY:
A randomized controlled trial was conducted with 100 critically ill pregnant women admitted to our hospital's obstetrics ICU between January 2023 and December 2024. Participants were allocated via random number table to either the control group receiving conventional multidisciplinary resuscitation care (n=50) or the observation group receiving the structured team model with shared decision-making (n=50). Comparative outcomes included resuscitation efficiency indicators (pre-hospital response time, intrahospital transport duration, emergency supply preparation time), complication rates, family psychological status measured by Hospital Anxiety and Depression Scale (HADS), and family satisfaction assessments

ELIGIBILITY:
Inclusion Criteria:

* Meeting diagnostic criteria for critical obstetric conditions:

  1. Amniotic fluid embolism
  2. Postpartum hemorrhage
  3. Emergency cesarean section was performed, etc
* Age ≥18 years
* Gestational age >20 weeks
* Patient's family/legal representative capable of normal communication and providing signed informed consent

Exclusion Criteria:

* Pre-existing primary hematologic disorders:
* Fetal congenital anomalies confirmed by prenatal imaging
* Active malignant tumors (except carcinoma in situ)
* Severe organ dysfunction:
* Altered mental status (GCS ≤12) or documented psychiatric disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Maternal mortality in critically ill women | 28 days postpartum
  The mortality of critically ill parturients during hospitalization and the number of deaths/total number of parturients were recorded.
Neonatal survival rate | Seven days after birth
  counting the survival of newborns within seven days after birth

SECONDARY OUTCOMES:
pre-hospital response time | 1 day
  The pre-hospital emergency response time was recorded
intrahospital transport duration | 1 day
  The intra-hospital transport time was recorded
emergency supply preparation time | 1 day
  The preparation time of first aid items was recorded
complication rates | 28 days postpartum
  Complications such as fever, infection and pelvic hematoma were recorded during the rescue period.
family psychological status measured | 28 days postpartum
  The Hospital Anxiety and Depression Scale (HADS) was used for evaluation, which consists of two subscales, including anxiety and depression, each with 7 items. The scale is scored on a 4-point scale, and the total score is 0-21. The higher the score, the more serious the anxiety or depression.
Satisfaction of family members | 28 days postpartum
  The Chinese version of critical care family satisfaction survey (CCFSS) was used for evaluation. The scale consisted of 5 dimensions and 20 items, including disease assurance, access to information, acceptance, support, and comfort. There were 4, 5, 3, 6, and 2 items in sequence, and a 5-point scale was used. The total score ranged from 20 to 100, with higher scores indicating higher family satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantong First People's Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
We may have further research, and we may not consider releasing the research data until the results are announced

REFERENCES:
- [Derived] Lu Y, Cai H, Chen L, Ni X, Ji J, Zhou Y, Liu Y, Jiang Y, Wang Y. Application of structured team model based on shared decision model in obstetrics and gynecology joint intensive care unit (ICU) rescue of critical care pregnant women: A randomized controlled trial. Medicine (Baltimore). 2025 Sep 5;104(36):e44430. doi: 10.1097/MD.0000000000044430. PMID 40922285